CLINICAL TRIAL: NCT02868346
Title: Improving the Diagnosis of Sexually Transmitted Infections in Emergency Rooms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-50; 2012-A01599-34 (Other: ANSM)
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Sexually Transmitted Infection
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients admitted for sexually transmitted infection (Experimental)
  Interventions: Other: Anal swab

INTERVENTIONS:
Other: Anal swab

SUMMARY:
A point-of-care laboratory (POC) was set at North Hospital, Marseille, France for the diagnosis in less than two hours of sexually transmitted infections caused by known pathogens, close to the reception of Emergency service. In this instance 30% of patients have no etiological diagnosis after the POC sexually infection transmitted tests .

Most sexually transmitted infections can be diagnosed from an anal swab which is not routinely performed. In this study, we suggest to test the hypothesis that anal swab in addition to the routine genital swab would increase by at least 5% the diagnosis capacity of sexually transmitted infections after the POC tests.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted for sexually transmitted infection in emergency room requiring a microbiological examination with a "Sexually Transmitted Infection POC kit"
* Patient who freely signed the informed consent form
* Patient affiliated to a social security regime

Exclusion criteria

* Pregnant or breastfeeding women
* Adult patient under guardianship
* Patient deprived with liberty under court order
* Patient refusing or unable to sign the informed consent form

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2013-03-29 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with a confirmed etiological diagnosis of sexually transmitted infection | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Catherine GEINDRE, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided